CLINICAL TRIAL: NCT06735040
Title: The Effect of Photobiomodulation Therapy on Fatigue and Behavioural Status in Patients With Hashimoto's Thyroiditis
Brief Title: Effect of Photobiomodulation Therapy in Patients With Hashimoto's Thyroiditis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Sümeyye TUNÇ, Assistant Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMU-FTR-ST-03
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Hashimoto Thyroiditis; Thyroiditis
Keywords: Anxiety; Depression; Fatigue; Photobiomodulation Therapy; Low Level Laser Therapy
MeSH Terms: conditions — Hashimoto Disease; Thyroiditis; Anxiety Disorders; Depression; Fatigue | interventions — Low-Level Light Therapy; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Randomised, sham-controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients in the groups did not have information with regard to which group they were included in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation Therapy Group (Active Comparator): All patients diagnosed with HT in the study were receiving LT4 treatment. In the PMBT group, in addition to thyroid hormone replacement therapy, a continuous wave GaAIAs type diode laser device (Intelect® Mobile Laser, Model No: 2779, Production Year: 2016; Chattanooga Group) was also applied to the thyroid gland in a 0.07 cm² treatment area. Continuous mode at 850 nm wavelength, 100 mW output power, 1.43 W/cm2 power density and 28.57 J/cm2 energy density (28.57 J/cm2 =100 Mw x 20 s/0.07) were used during the photobiomodulation therapy.
  Interventions: Other: Photobiomodulation Therapy
- Sham Group (Sham Comparator): In the sham PMBT group, the probe was placed similarly to the treatment group. The screen of the laser device was active; however, the energy was set to 0 J and the power to 0 Mw, and the same procedures were also performed.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Photobiomodulation Therapy — Before each treatment session, the borders of the thyroid gland were marked with ultrasound by an endocrinology specialist. Eight target points (superior, mediolateral, inferior borders of the right and left thyroid lobes, right and left side of the isthmus) were demarked with a surgical pen. PMBT was applied to the marked areas on the thyroid gland, which were approximately 1 cm apart from each other.
  Other Names: Low Level Laser Therapy
  Arms: Photobiomodulation Therapy Group
Other: Sham — In the sham PMBT group, the probe was placed similarly to the treatment group. The screen of the laser device was active; however, the energy was set to 0 J and the power to 0 Mw, and the same procedures were also performed.
  Arms: Sham Group

SUMMARY:
The standard lifelong treatment for Hashimoto's thyroiditis (HT), a chronic autoimmune disease, is levothyroxine (LT4) therapy. Despite LT4 replacement therapy, patients continue to experience persistent fatigue, deterioration in psychological and general well-being. Our study was conducted to investigate the effects of photobiomodulation therapy (PMBT) combined with LT4 replacement therapy on fatigue and behavioural status in patients with HT.

DETAILED DESCRIPTION:
Photobiomodulation therapy (PMBT) induces a wide range of molecular, cellular and tissue-based therapeutic effects through a biostimulation process by inducing a photochemical reaction in the cell. Some investigations show useful effects of this treatment with regard to thyroid function, autoimmunity and vascularisation in patients with Hashimoto's thyroiditis (HT). However, little is known about the efficacy of PMBT on neuromuscular symptoms and behavioural status. Therefore, in this study we aim to contribute the present literature on PMBT and to determine the clinical efficacy of PMBT. To the best of our knowledge, this study is the first paper to discuss the symptomatic efficacy of PMBT in patients with HT. Here, we investigate the effects of PMBT applied in combination with LT4 treatment on fatigue, sleep quality and behavioural status in people diagnosed with HT.

ELIGIBILITY:
Inclusion Criteria:

* The study included patients over the age of eighteen years who were diagnosed with HT by a specialist physician and followed up with LT4 treatment.

Exclusion Criteria:

* Exclusion criteria were acute infection, use of immunosuppressants, immunostimulants and drugs that interfere with the production, transport and metabolism of thyroid hormones (e.g. corticosteroids, lithium and amiodarone), thyroid nodules, tracheal stenosis, history of serious illness (e.g. cancer, ischaemic coronary artery disease, stroke, renal and liver failure), history of exposure to ionising radiation or neoplasia in the cervical region, malignancy and thyroid surgery; cancer, ischaemic coronary artery disease, stroke, renal and hepatic failure), history of exposure to ionising radiation or neoplasia in the cervical region, history of malignancy and thyroid surgery, hypothyroidism caused by postpartum thyroiditis, pregnancy and lactation, neurological and psychiatric disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Fatigue Level | 3 months
  Fatigue level in all patients was assessed by Fatigue Impact Scale (FIS) and Fatigue Severity Scale (FSS). The FIS is a forty-item scale indicating the consequences of fatigue on daily life such that it includes cognitive, physical and psychosocial subscales. The sum of the subscales ranges from 0 to 40 (physical and cognitive) and 0-80 (psychosocial); a higher score indicates a more severe impact of fatigue in daily life. FSS assesses the degree of physical fatigue over the past week and includes nine items. Patients indicate how much they agree or disagree with the statements for each item on a seven-point Likert scale. FSS scores ≥ 4.0 indicate clinically relevant fatigue.
Feeling of General Fatigue | 3 months
  General fatigue feeling of the individuals were evaluated by Visual Analogue Scale (VAS).Individuals were asked to mark their fatigue level on the scale. '0' means 'not tired at all' and '10'means 'very tired'.

SECONDARY OUTCOMES:
Sleep Quality | 3 months
  The Pittsburgh Sleep Quality Index (PSQI) was used to assess sleep quality based on participants' sleep experiences in the past week. The PSQI is a self-administered questionnaire that has been proven to be a valid and reliable tool for measuring sleep quality and quantity. The PSQI consists of a total of seven components and nineteen questions, including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication and daytime dysfunction. The sum of the seven dimensional components gives global scores ranging from 0 to 21, with higher scores indicating poorer sleep quality. Those having score above 5 are considered as to have "poor sleep quality" and those having score 5 and below are considered as to have "good sleep quality" .
Sleepiness | 3 months
  Epworth Sleepiness Scale (ESS) was used to assess sleepiness. The ESS is a short, easy-to-administer questionnaire that subjectively assesses daytime sleepiness. The probability of falling asleep in the eight-day condition is determined by a scoring from 0 to 3 (0=no chance of napping, 1=slight chance of napping, 2=moderate chance of napping, 3=high chance of napping). The ESS score is the sum of eight item scores and ranges from 0 to 24. Higher ESS scores indicate greater daytime sleepiness.
Anxiety | 3 months
  The inventory consists of twenty-one items describing subjective, somatic or panic-related anxiety symptoms, respectively. Self-reports are based on a four-point Likert scale ranging from "not at all" to "severe" regarding the experience of this symptom in the past month. Higher scores indicate more severe levels of anxiety.
Depression | 3 months
  The Beck Depression Inventory (BDI) is a twenty-one-item self-assessment scale that measures symptoms of depression. Each item is scored from 0 to 3; the total score ranges from 0 to 63. It was stated that those having scores as seventeen and above were in the group at risk of depression. Depression levels: 0-9, minimal; 10-16, mild; 17-29, moderate; 30-63, severe.

CONTACTS AND LOCATIONS:
Overall Officials: Şükriye Leyla ALTUNTAŞ, Study Director — Medipol University; Murat ATMACA, Study Chair — Medipol University
Locations (1):
- Sümeyye TUNÇ, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No